CLINICAL TRIAL: NCT06585111
Title: The Effect Of Individual Counseling Interventions Based On Health Action Process Approach Model On Breastfeeding Duration In Twin Pregnancies
Brief Title: Effect of Individual Counseling Interventions Based On Health Action Process Approach Model On Breastfeeding Duration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, ÇİĞDEM KÖPRÜLÜ, Specialist Nurse, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EGEU-SBF-CK-01
Record Dates: First submitted 2024-08-10; First posted 2024-09-05 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Breast Feeding
Keywords: Breas Feeding; Twins; Motivational Interviewing; Self Efficacy
MeSH Terms: conditions — Breast Feeding | interventions — Methods

STUDY DESIGN:
Intervention Model Description: The participants were divided into two groups: intervention and control groups. Interventions and follow-ups were carried out in six determined time periods.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breastfeeding Education (Experimental): Women in the intervention group received breastfeeding education through six motivational interviews based on the Health Action Process Approach (HAPA) Model (antenatal period 28-38 weeks, postpartum period 1-3 days, postpartum period 1-2 weeks, postpartum period 4-6 weeks, postpartum period 4th month, postpartum period 6th month).
  Interventions: Other: Intervention
- Control (No Intervention): The women in the control group received six follow-ups based on the Health Action Process Approach (HAPA) Model (antenatal period 28-38 weeks, postpartum period 1-3 days, postpartum period 1-2 weeks, postpartum period 4-6 weeks, postpartum period 4th month, postpartum period 6th month).

INTERVENTIONS:
Other: Intervention — In the first motivational interview, the "HAPA Model Prenatal Motivation Interview Questionnaire", the first part of the "Personal Information Form", the "Prenatal Breastfeeding Self-Efficacy Scale", and the "Breastfeeding Intention Scale for Pregnant Women Expecting Twins" were applied. A brochure on breastfeeding twin babies prepared by the researcher was distributed to women. In the second interview, the "HAPA Model Postpartum Motivation Interview Scale", the second part of which was the "Personal Information Form", "Breastfeeding Follow-up Form", "Breastfeeding Motivation Scale" and "Postpartum Breastfeeding Self-Efficacy Scale" were applied. In the third meeting, the "Breastfeeding Follow-up Form" was applied. "Breastfeeding Motivation Scale", "Postpartum Breastfeeding Self-Efficacy Scale" and "Breastfeeding Follow-up Form" were applied in the fourth and fifth interviews, and "Breastfeeding Follow-up Form" was applied in the sixth interview.
  Arms: Breastfeeding Education

SUMMARY:
The aim of this prospective, randomized controlled experimental clinical trial was to examine the effect of individual counseling interventions based on the Health Action Process Approach Model on breastfeeding duration in twin pregnancies. Women in the intervention group received breastfeeding education using motivational interviewing techniques, while women in the control group received routine clinical education and no intervention. Hypotheses of the study:

H1: Women who received individual intervention based on the SESY model have higher prenatal breastfeeding self-efficacy than the control group.

H2: Women who received individual intervention based on the SESY model have higher prenatal breastfeeding intentions than the control group.

H3: Postnatal breastfeeding self-efficacy of women who received individual intervention based on SESY model is higher than the control group.

H4: Breastfeeding motivation of women who received individual intervention based on the SESY model is higher than the control group.

H5: Women who received individual intervention based on the SESY model had higher rates of exclusive breastfeeding than the control group.

The women in the intervention group were given breastfeeding education with motivational interviewing techniques at 28-38 weeks of pregnancy in the prenatal period and 1-3 days, 1-2 weeks, 4-6 weeks, 4th month and 6th month in the postpartum period. The women in the control group did not receive any training by the researcher.

DETAILED DESCRIPTION:
Evaluate the effect of individual counseling interventions based on the Health Action Process Approach Model (HAPA) on breastfeeding duration in twin pregnancies.

A total of 34 women in the intervention group and 34 women in the control group were followed up six times at 28-38 weeks in the antenatal period and 1-3 days, 1-2 weeks, 4-6 weeks, 4th month and 6th month in the postpartum period. Personal Information Form, HAPA Model Antenatal Period Motivational Interview Questionnaire, HAPA Model Postpartum Period Motivational Interview Questionnaire, Prenatal Breastfeeding Self-Efficacy Scale, Breastfeeding Intention Scale in Pregnant Women Expecting Twins, Breastfeeding Follow-up Form, Breastfeeding Motivation Scale Turkish version, Postnatal Breastfeeding Self-Efficacy Scale were applied to the intervention group. In the control group, Personal Information Form, Prenatal Breastfeeding Self-Efficacy Scale, Breastfeeding Intention Scale in Pregnant Women Expecting Twins, Breastfeeding Follow-up Form, Breastfeeding Motivation Scale Turkish version, Postnatal Breastfeeding Self-Efficacy Scale were applied and they were followed up with routine clinical trainings.

ELIGIBILITY:
Inclusion Criteria:

* Who agreed to participate in the study,
* 18 years of age or older,
* Can speak and understand Turkish,
* Can read and write,
* Mothers whose breasts are suitable for breastfeeding
* Weeks between (28+0)-(37+6) of pregnancy

Exclusion Criteria:

* The baby has an anomaly in the mouth area
* The woman has language and communication problems
* The breasts are not suitable for breastfeeding (history of mastectomy surgery on both breasts)
* The mother or the baby is taking medication that prevents breastfeeding
* The woman has a previously diagnosed psychiatric disorder
* The mother does not plan to breastfeed her babies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Breastfeeding duration of twin babies until the sixth month postpartum after counseling | Postpartum 1-3 days, postpartum 1-2 weeks, postpartum 4-6 weeks, postpartum 4 months and postpartum 6 months
  The duration of breastfeeding the twins was measured using a breastfeeding follow-up form after the counseling intervention using motivational interviewing techniques. The breastfeeding follow-up form included questions about the number of breastfeedings in the last 24 hours and the mothers' formula feeding status. Mothers who breastfed 9-12 times were considered to have breastfed their babies sufficiently. Mothers who breastfed their babies 6 times or less did not breastfeed their babies enough. Babies of mothers who give formula to their babies are interpreted as not receiving enough breast milk.

SECONDARY OUTCOMES:
Duration of exclusive breastfeeding of twin babies after consultation until the sixth month after birth | postpartum 1-3 days, postpartum 1-2 weeks, postpartum 4-6 weeks, postpartum 4 months and postpartum 6 months
  The duration of breastfeeding the twins was measured using a breastfeeding follow-up form after the counseling intervention using motivational interviewing techniques. The breastfeeding follow-up form included questions about the number of breastfeedings in the last 24 hours and the mothers' formula feeding status. Mothers who breastfed 9-12 times were considered to have breastfed their babies sufficiently. Mothers who breastfed their babies 6 times or less did not breastfeed their babies enough. Babies of mothers who give formula to their babies are interpreted as not receiving enough breast milk.
Breastfeeding Intention Level | In the prenatal period between 28-38 weeks of gestation
  The breastfeeding intention level of mothers of twin babies was measured with the breastfeeding intention scale in the prenatal period.The scale is a 5-point Likert scale. Items are scored from strongly disagree 1 to strongly agree 5. A minimum of 7 and a maximum of 35 points can be obtained from the scale. The higher the total score obtained from the scale, the higher the breastfeeding intention of pregnant women expecting twins. The scale can be used in both primiparous and multiparous pregnant women from the 20th gestational week until delivery. The scale can be easily completed by literate individuals.
Prenatal Breastfeeding Self Efficacy Level | In the Prenatal period between 28-38 weeks of gestation
  The prenatal breastfeeding self-efficacy level of the mothers of twin babies was measured with the prenatal breastfeeding self-efficacy scale after breastfeeding training with motivational interviewing techniques. The scale consists of a total of 19 items and four subgroups. Each item of the scale is classified as "1=Not at all sure", "2=Slightly sure", 3=Quite sure", 4=Very sure", 5= Completely sure". It is graded on a 5-point Likert scale. The lowest score that can be obtained from the total scale is 19 and the highest score is 95. It is evaluated over the total score. The higher the score, the higher the perception of breastfeeding self-efficacy.
Postnatal Breastfeeding Self Efficacy Scale Level | Postpartum 1-3 days, postpartum 4-6 weeks, and postpartum 4th month.
  The postpartum breastfeeding self-efficacy levels of the mothers of twin babies were measured with the postnatal breastfeeding self-efficacy scale after breastfeeding training with motivational interviewing techniques. The Breastfeeding Self-Efficacy Scale developed by Dennis in 1999 consists of 33 items. Dennis developed the short form of the Breastfeeding Self-Efficacy Scale in 2003 by reducing it to 14 items. The Short Form Breastfeeding Self-Efficacy Scale is a 5-point Likert-type scale with 1= "I am never sure" and 5 = "I am always sure". The higher the score, the higher the breastfeeding self-efficacy.
Breastfeeding Motivation Level in Mothers of Twin Babies | 1-3 days postpartum, 4-6 weeks postpartum, and 4th month postpartum
  The level of breastfeeding motivation in mothers of twin babies was measured by motivational interviewing techniques and breastfeeding motivation scale after breastfeeding education. The scale consists of 24 items. The scale was adapted into Turkish by Mızrak and Özerdoğan in 2017. The scale consists of 6 sub-dimensions. These are; integrated regulation first sub-dimension 13,14,16,19,15,21,18,24,22,23, intrinsic motivation and identified regulation second sub-dimension 11,8,16,3,14.6,8,11,13, internalized regulation-social approval third sub-dimension 4,5, internalized regulation-social pressure fourth sub-dimension 7,9, external regulation-infant health fifth sub-dimension 2,12. and external regulation-additional benefits sixth sub-dimension 20,1,17,10. Scale items are graded from 1=strongly disagree to 4=strongly agree.

CONTACTS AND LOCATIONS:
Overall Officials: Oya Kavlak, Prof. Dr., Study Director — Ege University
Locations (1):
- Ege University, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Participant data will be shared with other researchers after the study is published (after 6 months).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Participant data will be shared with other researchers after the study is published (after 6 months).
Access Criteria: The national thesis center will make the thesis available to other researchers six months after approval.